CLINICAL TRIAL: NCT03115229
Title: The Effects of Protectıve Nursing Interventions on Reduction of Obesity Risk In University Students: Randomized Controlled Study
Brief Title: Obesity Intervention Program for University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Tuba Demirel, Selçuk University Coordinator of Scientific Research Projects, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 15102038
Record Dates: First submitted 2017-03-22; First posted 2017-04-14 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2017-03

CONDITIONS: Obesity
Keywords: Obesity; Overweight; Physical Activity; Nutrition; Nursing
MeSH Terms: conditions — Obesity; Overweight; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In the RCT, blindness was done in terms of data collectors and statistician. The data were collected by another investigator (assistant investigator) who did not know who was in the experiment and control group, and the data were recorded by the assistant investigator on the computer, without specifying the experiment and control group.
  Experimental and control groups were coded by an assistant investigator. Analysis of the data encoded by groups was done by a statistician.
  After the statistical analyzes were made and the research report was written, the assistant investigator explained the coding for the experiment and control group.
  In this way, data gathering, statistical analysis and reporting have been blinded.
  Note: Two assistant researchers received support from the research process. One of the assistant researcher is a coach who is a graduate of the Faculty of Sport Sciences other than Ph.D. Student of the Department of Public Health Nursing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group of the RCT was composed of 35 students randomly assigned to the control group who are BMI was between 25.0-29.9 or BMI was between 18.5-24.9 and they were in the risk group in terms of obesity according to the risk rating scales.
- Intervention Group (Experimental): The selected students were associated with obesity risk factors about obesity (owerveight or normal weight and they were in the risk group in terms of obesity according to the risk rating scales, and between 19-24 years old) and randomly assigned to the experimental group to Protective Nursing Interventions for Reduction Obesity Risk
  Interventions: Behavioral: Protective Nursing Interventions for Reduction Obesity Risk

INTERVENTIONS:
Behavioral: Protective Nursing Interventions for Reduction Obesity Risk — Applications for the experimental group for 11 weeks are grouped under three headings.
  These; Nutritional habits, practices for physical activity, and motivational messages sent via social media.
  Nutritional practices: Nutritional practices consist of group trainings, individual practices and collective events.
  Practices for physical activity: Group trainings, group exercises, individual exercises and collective activities. Physical activity was done for 3 days per week and 45-60 minutes every seans for 8 weeks. In addition, activities such as collective nature walks and cycling have been carried out Practices through social media: For physical activity and healthy eating; Motivational messages were sent twice a week for 11 weeks.
  Arms: Intervention Group

SUMMARY:
The aim of this study is to determine the effect of preventive nursing interventions, which consist of education / practices including of healthy eating and physical activity and motivational messages which sent through social media to reduce obesity risk in university students who in the risk group for obesity.

DETAILED DESCRIPTION:
This study has been conducted with University students in Turkey. The selected 70 students were associated with obesity risk factors about obesity (owerveight or normal weight and they were in the risk group in terms of obesity according to the risk rating scales, and between 19-24 years old) and randomly assigned to the experimental (35 students) and control group (35 students). Applications for the experimental group for 11 weeks about nutritional habits, practices for physical activity, and motivational messages sent via social media.

Primary Outcome Measure: Nutrition-Exercise Attitude Score, Nutrition-Exercise Behavior Score, Exercise Benefit / Obstacle Score. We used some scales for evaluate the primary outcomes (The Scale of Nutrition-Exercise Attitude-Behavior, The Scale of Exercise Benefit / Obstacle).

Bady Mass Index, Waist / Hip Ratio and Body fat percentage are secondary outcomes.

The data was calculated with SPSS package program.

ELIGIBILITY:
Inclusion Criteria:

* Preobezes between 25.0-29.9 BMI
* The BMI is 18.5-24.9 and who get above the average score (24-36 points high risk) from the "Risky Behavior Scale University Form: the subscale of nutritional habits
* The BMI is 18.5-24.9 and who get below the mean score (8-20 points high risk) from the Healthy Lifestyle Behavior Scale's subscale of Exercise

Exclusion Criteria:

* BMI below 18.5 and above 29.9
* Constantly regular drug users
* Those who have any health problems (who have had a heart attack, angioplasty or any surgical operation within 3 months, those with heart failure, those with metabolic disease, those with eating disorder, those with cancer, those with any psychological disease, Physically disabled)
* Those who are pregnant
* Those who have participated in any weight management program at least 2 months in advance and are still involved in the nutrition or physical activity program

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2016-03-07 (Actual); Study Completion 2016-05-27 (Actual)

PRIMARY OUTCOMES:
Nutrition-Exercise Attitude Score, Nutrition-Exercise Behavior Score, Exercise Benefit / Obstacle Score | Totaly: 11 weeks
  The Scale of Nutrition-Exercise Attitude-Behavior, The Scale of Exercise Benefit / Obstacle

SECONDARY OUTCOMES:
Bady Mass Index | Totaly: 11 weeks
  Weight/Height Ratio
Waist / Hip | Totaly: 11 weeks
  Waist / Hip Ratio
Body fat percentage | Totaly: 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Belgin Akın, Professor, Study Director — Selcuk University

IPD SHARING:
Plan to Share IPD: No